CLINICAL TRIAL: NCT05706181
Title: Home-based Heat Therapy to Improve Functional Capacity and Vascular Health in Older Adults
Brief Title: Heat Therapy, Functional Capacity, and Vascular Health in Older Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UNorthTexas
Record Dates: First submitted 2022-12-21; First posted 2023-01-31 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-01

CONDITIONS: Aging Well; Walking, Difficulty; Hyperemia
Keywords: Healthy aging; Functional capacity; Exercise hyperemia; Vascular function; heat therapy
MeSH Terms: conditions — Mobility Limitation; Hyperemia; Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: With the exception of a research nurse, all research personnel are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based heat therapy and functional capacity in older adults (Experimental): The investigators will determine the extent to which home-based leg heat therapy improves functional capacity in older adults. Functional capacity will be assessed before and after heat therapy or sham intervention via the 6-min walk test and the Short Physical Performance Battery.
  Interventions: Other: Home-based leg heat therapy; Other: Home-based sham therapy
- Home-based heat therapy and vascular function and exercise hyperemia in older adults (Experimental): The investigators will determine if home-based leg heat therapy improves vascular function and exercise hyperemia in the older adults of Aim 1. Using state-of-the-art techniques of skeletal muscle microdialysis and high-resolution duplex ultrasound, the investigators will pharmacodissect mechanisms of vascular function and exercise hyperemia before and after each intervention. The outcomes of Aim 2, while providing insight into the mechanisms whereby heat therapy improves functional capacity, should be considered independent of the outcomes of Aim 1 given that vascular health is a key independent, yet modifiable risk factor for cardiovascular morbidity and mortality.
  Interventions: Other: Home-based leg heat therapy; Other: Home-based sham therapy

INTERVENTIONS:
Other: Home-based leg heat therapy — Participants will be required to perform 8 weeks of leg heat therapy using water-perfused pants 4 times per week, with each session lasting 60 min. Skin temperature will be heated to about 40 °C. The pants heating system (consisting of pants and a water circulator/heater) can finely and uniformly control these designated skin temperatures. Participants will be randomly assigned to a group and provided with the pant heating system as well as a log book in which they are required to track the dates of each session. Participants will also measure their blood pressure and heart rate prior to, during, and immediately after each heating session using a portable oscillometric device provided by our laboratory.
Other: Home-based sham therapy — Participants will be required to perform 8 weeks of leg heat therapy using water-perfused pants 4 times per week, with each session lasting 60 min. Skin temperature will be heated to about 40 °C. The pants heating system (consisting of pants and a water circulator/heater) can finely and uniformly control these designated skin temperatures. Participants will be randomly assigned to a group and provided with the pant heating system as well as a log book in which they are required to track the dates of each session. Participants will also measure their blood pressure and heart rate prior to, during, and immediately after each heating session using a portable oscillometric device provided by our laboratory.

SUMMARY:
To test the hypothesis that home-based leg heat therapy improves functional capacity, vascular function, and exercise hyperemia in older adults.

DETAILED DESCRIPTION:
Chronic whole-body heating (i.e., heat therapy) has gained attention as a novel strategy to improve clinical and physiological outcomes in a number of populations. However, whole-body heat therapy is quite uncomfortable and may require trained personnel to ensure participant safety, especially for those more at risk for heat-related illness. Moreover, the applicability and acceptability of whole-body heat therapy are questionable as equipment cost is substantial and adherence will be low if individuals are required to travel if they cannot afford in-home therapy. Home-based leg heat therapy offers an opportunity to leverage the demonstrated benefits of whole-body heat therapy while managing safety and convenience.

The hypothesis will be addressed in the following Specific Aims:

Aim 1: Determine the extent to which home-based leg heat therapy improves functional capacity in older adults. Functional capacity will be assessed before and after heat therapy or sham intervention via the 6-min walk test and the Short Physical Performance Battery.

Aim 2: Determine if home-based leg heat therapy improves vascular function and exercise hyperemia in the older adults of Aim 1. Using state-of-the-art techniques of skeletal muscle microdialysis and high-resolution duplex ultrasound, the investigators will pharmacodissect mechanisms of vascular function and exercise hyperemia before and after each intervention. The outcomes of Aim 2, while providing insight into the mechanisms whereby heat therapy improves functional capacity, should be considered independent of the outcomes of Aim 1 given that vascular health is a key independent, yet modifiable risk factor for cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. 55 to 80 years of age
2. No tobacco/nicotine use within preceding 6 months (e.g., cigarettes, chewing tobacco, nicotine gum or patches, and vapor smoking)
3. Systolic blood pressure <140 mmHg; diastolic blood pressure <90 mmHg
4. Normal 12-lead ECG (reviewed by a physician)
5. Normal clinical results from a medical exam reviewed by a board-certified physician (e.g., General Health Questionnaire - see attached document)
6. Body mass index (BMI) <40 unless athletic/muscular build; calculation = body weight (kg)/height (m2)
7. Females Only: Post-menopausal

Exclusion Criteria:

1. Not meeting the age criteria
2. Body mass index (BMI) >40 unless athletic/muscular build; calculation = body weight (kg)/height (m2)
3. Use of tobacco or nicotine products within the last 6 months (tobacco cigarettes, chewing tobacco, nicotine patches or gum)
4. Not abstaining from the following 24 hours prior to the experimental session: exercise, alcoholic substances, prescription or non-prescription medications (unless cleared by the medical screener), dietary supplements, herbal medications, caffeinated substances (including chocolate, coffee, tea (iced or hot), caffeinated energy drinks, and sodas)
5. S who weigh less than 80 lbs
6. Use of prescription drugs, non-prescription drugs or herbal medicines known to alter vascular function unless cleared prior to the study
7. Use of anti-hypertensive medications
8. Use of beta blockers
9. Daily use of bronchodilators
10. Current use of anti-coagulant therapy
11. Current use of hormone replacement therapy (e.g., estrogen, testosterone)
12. Current diagnosis of cancer
13. Signs of overt cardio-metabolic abnormalities (e.g., uncontrolled diabetes - HbA1c >7.5, a resting systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg; abnormal 12-lead ECG)
14. History of cerebrovascular abnormalities (e.g., prior stroke, transient ischemic attacks, epilepsy, increased intracranial pressure)
15. Known history of atherosclerosis (i.e., plaque formation)
16. Autonomic dysfunction (e.g., Shy-Drager Syndrome, Bradbury-Eggleston syndrome, idiopathic orthostatic hypotension)
17. Respiratory illnesses (e.g., chronic asthma (including exercise-induced asthma), Chronic Obstructive Pulmonary Disease, Reactive Airway Disease). Note: subjects with exercised-induced asthma or who have had COVID-19 will be allowed to participate
18. History of anaphylaxis
19. Severe phobia of needles
20. History of alcohol or drug abuse which inhibits the participants ability to complete this study
21. Latex allergy
22. Known allergies or sensitivities to drugs used in the study (e.g., Lidocaine HCL, acetylcholine HCL, methacholine chloride, sodium nitroprusside, nitroglycerin, or related drugs)
23. Implanted electronic medical devices (e.g. cardiac pacemaker)
24. Tissue or skin abnormalities of the legs (e.g., infection, injury, open wound, ischemic tissue, phlebitis, active bleeding, neuropathy)
25. Tissue or skin abnormalities of the arm (e.g., unhealed or open wound or circulatory deficits)
26. Current Fever (oral temp >99.5 °F/ 37.5 °C) aa) Current use of PDE3 inhibitors (e.g., Viagra) or soluble guanylate cyclase (sGC) stimulators (e.g., riociguat), or unwillingness to withhold medication for 2 weeks prior to laboratory testing bb) Diagnosis of neurological disease or cognitive dysfunction cc) Cardiac surgery or cardiac events (e.g., coronary artery bypass graft surgery, myocardial infarction, heart failure) dd) Abnormal clotting, clots in deep veins in the legs or pelvis, or blood clots to the lungs ee) Individuals who have had mastectomies ff) History of methemoglobinemia

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | Before sham or heat therapy
  The distance, in meters, covered while walking for 6 minutes will be used to assess functional capacity.
6 minute walk test | After 8 weeks of heat therapy or sham
  The distance, in meters, covered while walking for 6 minutes will be used to assess functional capacity.
Macrovascular function | Before sham or heat therapy
  High-resolution duplex ultrasound will be used to assess vasodilation following a 5 minutes of leg ischemia. Vasodilation will calculated as the percent change in diameter of the superficial femoral that occurs following ischemia.
Macrovascular function | After 8 weeks of heat therapy or sham
  High-resolution duplex ultrasound will be used to assess vasodilation following a 5 minutes of leg ischemia. Vasodilation will calculated as the percent change in diameter of the superficial femoral that occurs following ischemia.
Microvascular function | Before sham or heat therapy
  The microdialysis technique will be used to delivery small amounts of acetylcholine or methacholine and sodium nitroprusside to the skeletal muscle of the thigh. Endothelial-dependent and endothelial-independent microvascular function can then be examined by assessing the increase in skeletal muscles blood flow during the infusion of acetylcholine/methacholine and sodium nitroprusside, respectively.
Microvascular function | After 8 weeks of heat therapy or sham
  The microdialysis technique will be used to delivery small amounts of acetylcholine or methacholine and sodium nitroprusside to the skeletal muscle of the thigh. Endothelial-dependent and endothelial-independent microvascular function can then be examined by assessing the increase in skeletal muscles blood flow during the infusion of acetylcholine/methacholine and sodium nitroprusside, respectively.
Blood flow response to exercise | Before sham or heat therapy
  High-resolution duplex ultrasound will be used to assess the change in blood flow during graded plantar flexion exercise.
Blood flow response to exercise | After 8 weeks of heat therapy or sham
  High-resolution duplex ultrasound will be used to assess the change in blood flow during graded plantar flexion exercise.

SECONDARY OUTCOMES:
Physical performance Battery | Before sham or heat therapy
  Likert scale-based scores will be tabulated from a side-by-side stand test, semi-tandem stand test, and a tandem stand test.
Physical performance Battery | After 8 weeks of heat therapy or sham
  Likert scale-based scores will be tabulated from a side-by-side stand test, semi-tandem stand test, and a tandem stand test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No